CLINICAL TRIAL: NCT02512172
Title: A Study of Using Epigenetic Modulators to Enhance Response to MK-3475 in Microsatellite Stable Advanced Colorectal Cancer
Brief Title: A Study of Enhancing Response to MK-3475 in Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: J1538; IRB00060125 (Other: JHMIRB)
Record Dates: First submitted 2015-07-02; First posted 2015-07-30 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — cc-486; Azacitidine; romidepsin; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oral CC-486 & MK-3475 (Experimental): Oral CC-486 300 mg days 1-14 or 21 every 28 days + IV MK-3475 200 mg days 1 and 15 every 28 days
  Interventions: Drug: Oral CC-486; Drug: MK-3475
- Romidepsin & MK-3475 (Experimental): Romidepsin 14 mg/m2 days 1, 8 and 15 + IV MK-3475 200 mg days 1 and 15 every 28 days
  Interventions: Drug: Romidepsin; Drug: MK-3475
- Oral CC-486 & Romidepsin & MK-3475 (Experimental): Oral CC-486 300 mg days 1-14 or 21 + romidepsin 7 mg/m2 (days 1, 8 and 15) + IV MK-3475 200 mg days 1 and 15 every 28 days.
  Interventions: Drug: Oral CC-486; Drug: Romidepsin; Drug: MK-3475

INTERVENTIONS:
Drug: Oral CC-486
  Other Names: oral azacitidine; oral aza
  Arms: Oral CC-486 & MK-3475; Oral CC-486 & Romidepsin & MK-3475
Drug: Romidepsin
  Other Names: Istodax
  Arms: Oral CC-486 & Romidepsin & MK-3475; Romidepsin & MK-3475
Drug: MK-3475
  Other Names: pembrolizumab

SUMMARY:
This study is being done to test the safety and effectiveness of the combination of intravenous (IV) romidepsin and/or oral 5-azacitidine with IV MK-3475 in people with microsatellite stable (MSS) advanced colorectal cancer.

DETAILED DESCRIPTION:
This study is being done to test the safety and effectiveness of the combination of intravenous (IV) romidepsin and/or oral CC-486 with IV MK-3475 in people with microsatellite stable advanced colorectal cancer.

People with advanced colorectal tumors that are microsatellite stable (MSS) may join this study. Tumors that are MSS positive are not deficient in repair of DNA.

This is a pilot study that will look at different ways of making MSS colorectal tumors sensitive to MK-3475 by giving 14 or 21 days of an epigenetic agent (oral CC-486 and/or romidepsin).

Participants will be randomly assigned (by chance, like drawing numbers from a hat) to one of three study drug combinations:

A. Oral CC-486 taken daily for 21 days (and later shortened to 14 days if there are side effects) and IV MK-3475 given every 2 weeks.

B. IV romidepsin given once weekly for 3 weeks and IV MK-3475 given every 2 weeks C. Oral CC-486 taken daily for 21 days (and later shortened to 14 days if there side effects) and IV romidepsin given every 2 weeks and IV MK-3475 given every 2 weeks.

Each arm is repeated every 28 days and will continue until the point that the study drug are no longer working. It will not be possible to cross over onto another arm if a participant's disease does not respond to the study drugs.

In this study investigators are looking for the following information:

* What effects, good and/or bad, the combination of oral CC-486 and/or romidepsin in combination with MK-3475 has on participants' cancer; and
* If the genetic and chemical make-up of participants' blood and tumor cells play a role in a response to oral CC-486 and/or romidepsin in combination with MK-3475.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically confirmed microsatellite stable metastatic colorectal cancer and have received at least one line of treatment for metastatic colorectal cancer including fluoropyrimidines, oxaliplatin and/or irinotecan
2. Be willing and able to provide written informed consent/assent for the trial
3. Be 18 years of age on day of signing informed consent
4. Have measurable disease
5. Have biopsiable disease. If biopsy is attempted and unsuccessful (the patient undergoes an invasive procedure), the patient may still be treated
6. Have a performance status of 0 or 1 on the ECOG Performance Scale at study entry
7. Demonstrate adequate organ function
8. Female subject of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication
9. Female subjects of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication
10. Male subjects must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
11. In patients with liver metastases, there should be <50% involvement of the liver.
12. Patients must have had < 3 prior therapies in the metastatic setting.

Exclusion Criteria:

1. Patients whose tumors have progressed at the first restaging during first line therapy
2. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
4. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered from adverse events due to agents administered more than 4 weeks earlier
5. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks (6 weeks for nitrosureas or mitomycin C) prior to study Day 1 or who has not recovered from adverse events due to a previously administered agent
6. Has a known additional malignancy that is progressing or requires active treatment
7. Has known central nervous system (CNS) metastases and/or carcinomatous meningitis
8. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
9. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
10. Has an active infection requiring systemic therapy.
11. Any clinical or radiological ascites or pleural effusions
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX-40, anti-CD40, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways). Prior therapies with other immunomodulatory agents must be reviewed by the PI and may be cause for ineligibility
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
17. Has known active Hepatitis B or Hepatitis C
18. Has received a live vaccine within 30 days prior to the first dose of trial treatment
19. Any known cardiac abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Degree of change in tumor infiltrating lymphocytes | 1 year
  Change in the number of CD8+ TILs and/or the ratio of CD8+/CD4+ TILs in tumors pre- and post- treatment.
Number of Patients Experiencing a DLT (dose-limiting toxicity) as defined by NCI CTCAE v4.0 | 5 years
  Adverse events are defined by NCI CTCAE v4.0. The DLT observation period is one cycle (28 days).

SECONDARY OUTCOMES:
Immune-related Progression-free Survival (irPFS) at 20 weeks | 20 weeks
  irPFS rate is defined as the percentage of patients with disease progression (irPD or relapse from irCR as assessed using irRC criteria) or death due to any cause at 20 weeks. Per irRC criteria, Complete Response (irCR) is the disappearance of all target lesions, Partial Response (irPR) is a decrease in tumor burden by 50% or greater by a consecutive assessment at least 4 weeks after first documentation, Stable Disease (irSD) is the failure to meet criteria for irCR or irPR (in absence of irPD), Progressive Disease (irPD) is at least 25% increase in tumor burden relative to nadir. Estimation based on the Kaplan-Meier curve.
Overall Survival (OS) | 4 years
  OS will be measured from date of first dose until death or end of followup (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States